CLINICAL TRIAL: NCT00269126
Title: See Detailed Description
Brief Title: Clinical Evaluation Of GW815SF For Chronic Obstructive Pulmonary Disease (Chronic Bronchitis, Emphysema)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SCO100646
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2012-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Chronic Bronchitis; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol combination DISKUS
Drug: salmeterol xinafoate
  Other Names: fluticasone propionate/salmeterol combination DISKUS

SUMMARY:
This study compares the effect of two medicines on COPD (Chronic Obstructive Pulmonary Disease). This study will last up to 18 weeks, and subjects will visit the clinic 5 times. Subjects will be given breathing tests, and will record their breathing symptoms daily on diary cards.

DETAILED DESCRIPTION:
Clinical Evaluation of GW815SF for Chronic Obstructive Pulmonary Disease (Chronic Bronchitis, Emphysema) "Assessment of the Effect of Addition of Fluticasone Dipropionate to Salmeterol Xinafoate 50µg after Switching under Double-blinded conditions to GW815SF 50/250µg in Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD.

Exclusion criteria:

* Diagnosis of asthma or an uncontrolled medical condition or respiratory disorder other than COPD.
* Other inclusion and exclusion criteria will be evaluated at the first study visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pre-dose FEV1 at 4 weeks after starting medication of GW815SF 50/250µg

SECONDARY OUTCOMES:
Change in morning PEF
Changes in pre-dose FVC, V50, V25
Use of rescue medication
Changes in symptom scores

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Kyoto, Japan
- GSK Investigational Site